CLINICAL TRIAL: NCT03267472
Title: the Genitourinary Fistula Experience in Upper Egypt
Brief Title: Pattern of Genitourinary Fistula in Upper Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AHMED FARAHAT HASSAN, ahmed farahat hassan, Assiut University
Other Study IDs: genitourinary fistula
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the pattern of genitourinary fistula in upper egypt

DETAILED DESCRIPTION:
A genitourinary fistula is defined as an abnormal communication between the urinary (ureters, bladder, urethra) and the genital (uterus, cervix, vagina) systems.

The true incidence of genitourinary fistula is unknown. Uro-genital fistulas are a great challenge for women in developing countries.

The new classification of genitourinary fistula divides genitourinary fistulae into four main types, depending on the distance of the distal edge of the fistula from the external urinary meatus. These four types are further subclassified by the size of the fistula, extent of associated scarring, vaginal length or special considerations:

Type 1: Distal edge of fistula > 3.5 cm from external urinary meatus Type 2: Distal edge of fistula 2.5-3.5 cm from external urinary meatus Type 3: Distal edge of fistula 1.5 - < 2.5 cm from external urinary meatus

ELIGIBILITY:
Inclusion Criteria:

- any female with genitourinary fistula

Exclusion Criteria:

* no

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: A genitourinary fistula is defined as an abnormal communication between the urinary (ureters, bladder, urethra) and the genital (uterus, cervix, vagina) systems.
  The true incidence of genitourinary fistula is unknown. Uro-genital fistulas are a great challenge for women in developing countries. The new classification of genitourinary fistula divides genitourinary fistulae into four main types, depending on the distance of the distal edge of the fistula from the external urinary meatus.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2017-10-20 (Estimated); Study Completion 2017-10-20 (Estimated)

PRIMARY OUTCOMES:
prevalence of genitourinary fistula in upper egypt | 5 years
  to detect how many numbers of cases of genitourinary fistula in upper egypt .